CLINICAL TRIAL: NCT01406873
Title: A Randomized, Placebo Controlled, Clinical Efficacy Trial of Mexiletine for Myotonic Dystrophy Type-1 (DM1)
Brief Title: Clinical Efficacy Trial of Mexiletine for Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Chad Heatwole, Associate Professor of Neurology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3716; Funding Source: FDA/OOPD (Other Grant/Funding Number: R01FD003716)
Record Dates: First submitted 2011-07-20; First posted 2011-08-01 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Myotonic Dystrophy
Keywords: Myotonic Dystrophy; Myotonic Dystrophy Type 1 (DM1); Muscular Dystrophy; Mexiletine
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophies | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mexiletine (Active Comparator): 20 subjects will be randomized (assigned) to receive Mexiletine. Mexiletine is available on the market for the treatment of cardiac arrhythmias, but it is not currently approved for the treatment of myotonia or myotonic dystrophy.
  Interventions: Drug: Mexiletine
- Sugar pill (Placebo Comparator): 20 subjects will be randomized (assigned) to receive placebo (sugar pill). This control group is necessary to definitely establish the antimyotonic efficacy and safety of mexiletine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine — 150 mg/kg Mexiletine capsules taken by mouth, three times daily for 6 months
  Other Names: Generic name: mexiletine hydrochloride
  Arms: Mexiletine
Drug: Placebo — 150 mg/kg placebo capsules taken by mouth, three times daily for 6 months
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to investigate the effects of mexiletine treatment for 6 months on ambulation, myotonia, muscle function and strength, pain, gastrointestinal functioning, cardiac conduction, and quality of life in myotonic dystrophy type 1 (DM1).

DETAILED DESCRIPTION:
This study will provide data on the long term (6 months) safety and efficacy of mexiletine in:

* improving the distance participants are able to walk in six minutes;
* reducing myotonia;
* improving muscle strength;
* increasing lean muscle mass;
* decreasing musculoskeletal pain;
* improving gastrointestinal function and swallowing);
* improving functional abilities;
* decreasing cardiac arrhythmias; and
* improving disease-specific health related quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of DM1, confirmed by DM1 genetic mutation
* Ability to walk 30 feet (assistance with cane and/or leg bracing permitted)
* Presence of grip myotonia

Exclusion Criteria:

* Congenital DM1
* Treatment with Mexiletine within past 8 weeks
* Second or third degree heart block, atrial flutter, atrial fibrillation, ventricular arrhythmias, or is receiving medication for treatment of a cardiac arrhythmia
* Receiving another antimyotonia drug
* Liver or kidney disease requiring ongoing treatment
* Has a seizure disorder
* Is pregnant or lactating
* Had severe depression within 3 months or a history of suicide ideation
* Has any one of the following medical conditions: uncontrolled diabetes mellitus, congestive heart failure, symptomatic cardiomyopathy, symptomatic coronary artery disease, cancer (other than skin cancer) less than five years previously, multiple sclerosis, or other serious medical illness.
* Drug or alcohol abuse within 3 months
* Coexistence of another neuromuscular disease
* Is unable to give informed consent
* Severe arthritis or other medical condition (besides DM1) that would significantly impact ambulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Moxley, III, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Department of Neurology, Rochester, New York, United States

REFERENCES:
- [Background] Logigian EL, Martens WB, Moxley RT 4th, McDermott MP, Dilek N, Wiegner AW, Pearson AT, Barbieri CA, Annis CL, Thornton CA, Moxley RT 3rd. Mexiletine is an effective antimyotonia treatment in myotonic dystrophy type 1. Neurology. 2010 May 4;74(18):1441-8. doi: 10.1212/WNL.0b013e3181dc1a3a. PMID 20439846
- [Background] Moxley RT 3rd, Logigian EL, Martens WB, Annis CL, Pandya S, Moxley RT 4th, Barbieri CA, Dilek N, Wiegner AW, Thornton CA. Computerized hand grip myometry reliably measures myotonia and muscle strength in myotonic dystrophy (DM1). Muscle Nerve. 2007 Sep;36(3):320-8. doi: 10.1002/mus.20822. PMID 17587223

RESULTS

PARTICIPANT FLOW:
Groups:
- Mexiletine: This group received 150 mg/kg Mexiletine capsules taken by mouth, three times daily for 6 months
- Placebo: This group received 150 mg/kg placebo capsules taken by mouth, three times daily for 6 months
Period: Overall Study
Arm/Group | Mexiletine | Placebo
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mexiletine | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.05 (11.54) | 38.14 (9.78) | 40.10 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Ambulation Using the 6 Minute Walk Distance
Description: During this assessment, participants were asked to walk as far as they could back and forth on a fixed 20 meter route for 6 minutes. The total distance walked during the 6 minutes was recorded in meters. Change from baseline was defined as the difference between the average 6 minute walk distance at baseline and the average 6 minute walk distance at 6 months.
Time Frame: Baseline to 6 months
Population: Intent to Treat (ITT) population was defined as all participants who were randomized to the study, received at least one dose of study medication and have post-baseline efficacy assessment. Follow-up data was not collected on one participant in the mexiletine arm due to a broken foot.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Mexiletine: Mean Change from Baseline in Ambulation using the 6 Minute Walk Test in Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Mean Change from Baseline in Ambulation using the 6 Minute Walk Test in Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 19 | 20
Meters | 17.44 (39.84) | 7.25 (38.93)

2. Secondary Outcome: Percentage of Participants That Had a Dose Reduction or a Study Drug Withdrawal or Suspension Over 6 Months
Description: Adverse events were monitored at the three in-person evaluations (Months 0, 3, and 6), at telephone evaluations every 2 weeks, and via patient-completed side effect diaries. The study investigators and safety monitoring committee reviewed adverse events and made decisions regarding drug withdrawals, suspensions, and dose reductions as needed.
Time Frame: 6 months
Population: Intent to Treat (ITT) population was defined as all participants who were randomized to the study, received at least one dose of study medication and have post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Mexiletine: Percentage of Participants that had a dose Reduction or a Study Drug Withdrawal or Suspension for Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Percentage of Participants that had a dose Reduction or a Study Drug Withdrawal or Suspension for Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Study Drug Withdrawal | 2 | 0
  Study Drug Dose Reduction | 1 | 0
  Study Drug Temporary Suspension | 1 | 0

3. Secondary Outcome: Mean Change From Baseline in Quantitative Measure of Hand Grip Myotonia
Description: Relaxation time of the long finger flexor muscles of the right hand after a maximum voluntary isometric contraction performed in a standardized fixed position of the right arm elbow/wrist/hand. Relaxation time for this measurement is defined as the time to relax from 90% to 5% of the maximum isometric force of contraction of the hand (the first of 6 serial contractions averaged over two consecutive trials performed 10 minutes apart).
Time Frame: Baseline to 6 months
Population: Intent to Treat (ITT) population was defined as all participants who were randomized to the study, received at least one dose of study medication, and have post-baseline efficacy assessment at 6 months. Data was not analyzable on 3 people in the placebo arm.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Mexiletine: Mean Change from Baseline in Quantitative Measure of Hand Grip Myotonia for Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Mean Change from Baseline in Quantitative Measure of Hand Grip Myotonia for Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 20 | 17
Seconds | -1.01 (1.78) | 0.43 (1.53)
Statistical Analysis 1: Comparison: Mexiletine vs Placebo; Test type: Superiority; p < 0.01, ANCOVA

4. Secondary Outcome: Mean Change From Baseline in Manual Muscle Testing (MMT) Score
Description: Manual muscle testing was performed on 26 muscle groups (shoulder abductors, elbow flexors, wrist flexors, wrist extensors, hip flexors, knee extensors, hip extensors, knee flexors, hip abductors, elbow extensors, ankle dorsiflexors, and plantar flexors on the right and left plus neck extensor and neck flexors). The muscles were tested in various positions including sitting, supine, prone, and side lying and each graded on a modification of the Medical Research Council (MRC) scale of 0 to 5 (5 representing normal strength). Average MMT score is derived by averaging the individual MMT scores across the 26 individual muscles.
Time Frame: Baseline to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Mexiletine: Mean Change from Baseline in Manual Muscle Testing (MMT) Score for Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Mean Change from Baseline in Manual Muscle Testing (MMT) Score for Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 20 | 20
Units on a scale | 0.05 (0.23) | -0.06 (0.12)

5. Secondary Outcome: Mean Change From Baseline in PR, QRS, and QTc Intervals, and Average Minimum Heart Rate (HR) Via Electrocardiogram (ECG) Monitoring
Description: PR, QRS, and QTc intervals as well as average minimum heart rate (HR) were obtained through standard 12 lead electrocardiograms (ECGs). Values were computer generated and verified by the study investigator and study cardiologist.
Time Frame: Baseline to 6 Months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 20 | 20
Milliseconds
  PR Interval: number analyzed (Participants) | 20 | 18
  PR Interval | 11.35 (38.08) | 8.89 (13.20)
  QRS Interval | 0.70 (11.50) | 1.00 (6.37)
  QTc Interval | -4.40 (23.37) | -1.55 (14.75)
  Average Minimum Heart Rate | 0.65 (4.57) | -0.25 (5.72)

6. Secondary Outcome: Mean Change From Baseline in Patient-Reported Disease Burden and Quality of Life
Description: * The Myotonic Dystrophy Health Index (MDHI) is a validated disease-specific measure of patient-reported disease burden. The MDHI total score is a weighted average derived from 17 subscales. MDHI total scores range form 0-100 with 0 representing no patient-reported disease burden and 100 representing the most severe patient-reported disease burden.
  * The Individualized Neuromuscular Quality of Life Questionnaire (INQoL) is a measure of quality of life in neuromuscular disease. The INQoL summary score is a weighted average made up of 5 sub-domains. Scores range from 0-100, and can be interpreted as the percent of maximal detrimental impact on quality of life with higher scores indicating more detrimental impact.
  * The 36-Item Short Form Survey (SF-36) is a generic measure of quality of life across 8 domains. Two summary metrics are produced from the 8 domains, ranging from 0-100% with lower scores representing worse levels of functioning.
Time Frame: Baseline to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Mexiletine: Mean Change from Baseline in Patient-Reported Disease Burden and Quality of Life for Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Mean Change from Baseline in Patient-Reported Disease Burden and Quality of Life for Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
Number analyzed (Participants) | 20 | 20
Units on a scale
  INQoL | 5.11 (14.80) | 2.33 (12.84)
  MDHI | 0.01 (7.75) | -1.10 (10.02)
  SF-36 Physical Component Summary: number analyzed (Participants) | 20 | 19
  SF-36 Physical Component Summary | -1.73 (7.12) | -1.35 (7.22)
  SF-36 Mental Component Summary: number analyzed (Participants) | 20 | 19
  SF-36 Mental Component Summary | -0.62 (9.01) | -0.79 (9.22)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 7 months. This period included 6 months (starting from randomization) on study drug (mexiletine vs. placebo) and 1 month post discontinuation of study drug.
Description: 2 subjects experienced study related AEs prior to randomization; both were in the mexiletine arm and both AEs were 'Skin and subcutaneous tissue disorders - Other, rash' and related to study procedures (where Holter monitor electrodes were placed). They are not included in the AE data displayed.
Groups:
- Mexiletine: Adverse Events for Patients who Received Mexiletine (150 mg/kg capsules taken by mouth, three times daily for 6 months)
- Placebo: Adverse Events for Patients who Received Placebo (150 mg/kg capsules taken by mouth, three times daily for 6 months)
Arm/Group | Mexiletine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 21/21 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine (N=21) | Placebo (N=21)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine (N=21) | Placebo (N=21)
Cardiac disorders - Other, increased PVCs (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (2) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, gastric distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 5 (5)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 12 (21) | 15 (28)
Pain (General disorders) | 3 (3) | 1 (3)
Hepatobiliary disorders - Other, elevated GGT (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, elevated eosinophils (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, cut finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, tendinitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, wrist sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, extreme thirst (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Musculoskeletal and connective tissue disorder - Other, heel spur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (7)
Nervous system disorders - Other, idiopathic transient brain brainstem dysfuncti (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, imbalance (Nervous system disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, numbness (Nervous system disorders) | 3 (3) | 0 (0)
Nervous system disorders - Other, transient lack of focus (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (2)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Renal and urinary disorders - Other, bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, uterine fibroid (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, bumps on face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, hair thinning (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, cataract surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, gum surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Surgical and medical procedures - Other, laser eye surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, mole removal (Surgical and medical procedures) | 1 (2) | 0 (0)
Surgical and medical procedures - Other, molluscum removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, root canal (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, tubal ligation (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT01406873/Prot_SAP_000.pdf